CLINICAL TRIAL: NCT03264781
Title: The Effect of Cyclofem® for the Treatment of Irregular Uterine Bleeding in Implant Contraceptive Users; a Randomized Controlled Trial
Brief Title: The Effect of Cyclofem® for the Treatment of Irregular Uterine Bleeding in Implant Contraceptive Users
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OBCU
Record Dates: First submitted 2017-06-06; First posted 2017-08-29 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Uterine Bleeding
Keywords: Cyclofem®; Implant; Jadelle; Implanon; irregular uterine bleeding; randomized controlled trial
MeSH Terms: conditions — Uterine Hemorrhage; Menstruation Disturbances | interventions — CycloProvera; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Cyclofem group (Experimental): Medroxyprogesterone Acetate 25 mg plus Estradiol Cypionate 5 mg (Cyclofem®) 0.5 ml IM injection single dose
  Interventions: Drug: Cyclofem
- Placebo group (Placebo Comparator): normal saline 0.5 ml IM single dose
  Interventions: Drug: Cyclofem

INTERVENTIONS:
Drug: Cyclofem — Intramuscularly injection 0.5 ml of Cyclofem or placebo
  Other Names: Questionnaire and Menstrual record chart

SUMMARY:
The purpose of this study is to determine that once-a-month injectable contraceptive( Cyclofem® ) has the effect on treatment of irregular uterine bleeding in implant contraceptive users or not.

DETAILED DESCRIPTION:
Stratified randomization Implanon and Jadelle group were done using block randomization. The participants and investigators were blinded to treatment allocation, using drug coding that not revealed until the end of study. Research assistants and nurse who did not have involve in analyses data would follow the recruitment criteria and drug injection follow the code of drug.

All participants were collected demographic data, medical history, obstetrical and gynecological history, bleeding pattern before enrollment. Then physical exam and pelvic examination were performed for all participants. Participants received single dose intramuscular injection of Cyclofem® 0.5 ml or normal saline 0.5 ml as placebo on that day of recruitment to the study. Daily record of bleeding, spotting and side effect was done on record form.

ELIGIBILITY:
Inclusion Criteria:

* Implant (Jadelle or Implanon) inserted before enrollment with the symptom of bleeding disturbances for eight or more continuous days or a current bleeding-free interval of 15 days or less
* Regular menstruation at least 1 cycle before the usage of implant contraceptive
* Willingness to participate in a placebo-controlled study and ability to keep an accurate daily menstrual record
* No gynecological or serious medical diseases

Exclusion Criteria:

* Contraindication to estrogen or progesterone use such as

  * breast cancer
  * Liver cancer or tumor
  * Uncontrolled blood pressure (BP ≥160/100 mmHg )
  * History of atherosclerosis, vascular disease and high risk for VIE
  * History of ischemic stroke
  * Coagulopathy
  * Uncontrolled diabetes mellitus and complication
  * Cirrhosis
  * SLE with antiphospholipid positive
  * History of migraine with aura or age of 35 years old or more than with history of migraine non-aura
  * Age of 35 years old or more than with history of smoking more than 15 cigarettes per day
  * Postpartum 6 weeks
  * Plan for surgery procedure that need immobilization after surgery
* Previous treatment for 3 months before enrollment
* Allergic to drug component of Cyclofem® ( Medroxyprogesterone acetate , Estradiol cypionate)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects that bleeding stopped after treatment with Cyclofem or placebo | 12 weeks
  Menstrual record chart was using to record bleeding/spotting days

SECONDARY OUTCOMES:
Number of days that bleeding stopped between Cyclofem® and placebo for the treatment of irregular uterine bleeding in implant contraceptive users | 12 weeks
  Menstrual record chart was using to record bleeding/spotting days
Side effect of Cyclofem® for the treatment of irregular uterine bleeding in implant contraceptive users | 12 weeks
  Questionnaire was using to record adverse effect during follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Nitisa Tapanwong, MD, Principal Investigator — Department of Obstetrics and Gynecology of King Chulalongkorn Memorial Hospital
Locations (1):
- Chulalongkorn Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No